CLINICAL TRIAL: NCT01737554
Title: Catheter Resistance Monitoring to Predict Catheter-Associated Adverse Events in Children and Adolescents: A Feasibility Study
Brief Title: Catheter Resistance Monitoring to Predict Catheter-Associated Adverse Events in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CARMA
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Cancer; Hematologic Disorders
Keywords: Central venous access device; Catheter resistance monitoring
MeSH Terms: conditions — Neoplasms; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Participants include children with cancer and hematologic disorders who, as part of their standard clinical care, have a central venous access device (CVAD) used for infusion, withdrawal of blood, or hemodynamic monitoring.
  Intervention: Catheter resistance monitoring
  Interventions: Other: Catheter Resistance Monitoring

INTERVENTIONS:
Other: Catheter Resistance Monitoring — Weekly measurement of resistance to flow in the lumen(s) of a CVAD with the commercially available Alaris® Syringe Module IV pump. The aim is to identify an increase in resistance greater than normal variation. Inline pressure measurements will be recorded at multiple flow-rates and resistance will be estimated from the gradient of the pressure-flow curve.
  Other Names: CRM

SUMMARY:
Catheter occlusion and dysfunction are common complications of central venous access device (CVAD) use in children with cancer and hematologic disorders. These events can lead to interruption of therapy and may require device removal and replacement. Attempts to clear occlusion can cause device fracture.

There is a clear link between catheter occlusion and other serious complications including bloodstream infection and intravascular thrombosis.

There is evidence that catheter occlusion or dysfunction may be preceded by subclinical catheter narrowing, which could be detected by accurate measurement of catheter resistance.

This study aims to observe and describe the feasibility and results of catheter resistance monitoring (CRM) over time with the aim of prospectively identifying patients at high risk of catheter occlusion.

If CRM is feasible and proves to be sensitive and specific, it could provide an opportunity for preemptive therapy to prevent occlusion, which might also prevent bloodstream infection or thrombosis.

DETAILED DESCRIPTION:
Weekly measurement of catheter resistance will be determined using the Alaris® Syringe Module (Carefusion Inc., San Diego, USA), a commercially available, FDA-approved intravenous (IV) pump which is able to deliver accurate flow-rates and obtain accurate pressure measurements. The inline pressure will be measured at multiple flow-rates and resistance will be estimated from the gradient of the pressure-flow curve.

Primary Objective

* To describe the feasibility of weekly CRM in children and adolescents treated at St. Jude.

Secondary Objectives

* To describe patient and caregiver adherence with weekly CRM in children and adolescents treated at St. Jude.
* To explore the correlation between results of CRM and catheter occlusion or dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment for any disease at St. Jude Children's Research Hospital (SJCRH).
* Age ≥5 years to <25 years.
* Participant is using either a single or double lumen tunneled CVAD (ports will not be eligible) as part of standard clinical care.
* Participant anticipates being present weekly at SJCRH for at least 12 weeks

Exclusion Criteria:

* Plan to remove CVAD within 12 weeks.
* Expected survival less than 12 weeks
* Past enrollment in the CaRMA study or past catheter resistance monitoring

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be drawn from current St. Jude patients who have a central venous access device already in place as part of their standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of attended CRM visits which produce usable resistance data for all lumens of the CVAD | Weekly for 12 weeks from study entry or until discontinuation of CRM, whichever is shorter
  To describe the feasibility of CRM in children and adolescents treated at St. Jude, the proportion of attended CRM visits which produce usable resistance data for all lumens of the CVAD will be recorded for each participant, and summary statistics, including median, range and standard deviation will be reported for the study population.

SECONDARY OUTCOMES:
Attendance at each planned CRM visit | Weekly for 12 weeks or until discontinuation of CRM for a prescribed reason, whichever is shorter
  To describe patient and caregiver adherence with weekly CRM in children and adolescents treated at St. Jude, attendance at each planned CRM visit will be recorded. Summary statistics for proportion of planned visits attended for each participant, including median, range and standard deviation will be reported for the study population.
The relationship between CRM results and occlusion or dysfunction | Up to 15 weeks
  To explore the correlation between the results of CRM and catheter occlusion or dysfunction in children and adolescents, the relationship between CRM results and occlusion or dysfunction will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wolf, MBBS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Wolf J, Tang L, Rubnitz JE, Brennan RC, Shook DR, Stokes DC, Monagle P, Curtis N, Worth LJ, Allison K, Sun Y, Flynn PM. Monitoring Central Venous Catheter Resistance to Predict Imminent Occlusion: A Prospective Pilot Study. PLoS One. 2015 Aug 31;10(8):e0135904. doi: 10.1371/journal.pone.0135904. eCollection 2015. PMID 26322512
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols